CLINICAL TRIAL: NCT05640531
Title: Phase-I, Double-blind, Randomized, Placebo-controlled Single Center Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses of Intravenous WCK 771 in Adult Healthy Human Volunteers
Brief Title: Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses of Intravenous WCK 771
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: WCK771/P-I/MD/08
Record Dates: First submitted 2021-04-30; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Bioavailability

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- WCK 771 (Experimental): WCK 771 600mg, 800mg, and 1000mg WCK 771 BID. Dosage form : IV Infusion
  Interventions: Drug: WCK 771 IV Infusion
- Placebo infusion (Placebo Comparator): Matching Placebo administered as IV infusion
  Interventions: Other: Placebo IV Infusion

INTERVENTIONS:
Drug: WCK 771 IV Infusion — subjects will receive intravenous infusion of WCK 771
  Arms: WCK 771
Other: Placebo IV Infusion — subjects will receive matching placebo intravenous infusion
  Arms: Placebo infusion

SUMMARY:
The present study is planned to assess the safety and pharmacokinetic profile in normal healthy subjects in US for WCK 771 with doses ranging from 600 mg to 1000 mg BID for 5 days. In the proposed Phase I MAD study, a subject will be administered 600mg, 800mg, and 1000mg WCK 771 BID for 5 days (Ten doses) or an identical placebo as intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

* Have a Body Mass Index (BMI) between 18 and 32 (both inclusive), calculated as weight in kg/height in m2
* Have no significant diseases or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations and ECG recordings

Exclusion Criteria:

* Known hypersensitivity or idiosyncratic reaction to quinolones or any other related drugs
* Any history or evidence of disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system
* Use of any prescription drug within 14 days prior to start of the study (check-in) and nonprescription drug within 7 days prior to start of study (check-in)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2012-02-07 (Actual); Study Completion 2012-06-27 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety & tolerability of multiple doses of WCK 771 | Day 12
  By monitoring the adverse events reported
To evaluate the pharmacokinetics of multiple doses of WCK 771 | Day 5
  Measuring Cmax Maximum observed plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Ashima Bhatia, MD, Study Director — Wockhardt Ltd
Locations (1):
- PPD Phase I Clinic, 7551 Metro Center Drive, Suite 200, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No